CLINICAL TRIAL: NCT05716217
Title: Can Training of the Armsy Reduce Pain When Inserting a Peripheral Venous Catheter, and How is it Experienced That There Can be Challenges With Vein Status for Patients in Cytostatic Treatment?
Brief Title: Training of Arms to Reduce Pain With Peripheral Venous Catheter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in provision of chemotherapy have made it impossible to recruit patients according to the protocol
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vein-project
Record Dates: First submitted 2023-01-25; First posted 2023-02-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pain; Cancer; Veins
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Intervention Model Description: One group is randomly assigned to an 8-week daily arm training program. The other group receives normal care
Who Masked: Care Provider
Masking Description: The anaesthesia nurses inserting PVCs and registering data are blinded to the participants' study allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental)
  Interventions: Other: Arm training
- Normal care (No Intervention)

INTERVENTIONS:
Other: Arm training — Daily arm training program
  Arms: Training group

SUMMARY:
Female patients undergoing chemotherapy for breast cancer often experience pain and discomfort when a peripheral venous catheter is inserted.

This randomized, controlled trial investigates whether there is a difference in the degree of pain during PVC insertion in patients who exercise their arms, and whether exercise improves vein status.

Participation involves:

* Everyone must have had their peripheral venous catheter (PVC) inserted at least five times in the DROP-IN, which is an outpatient clinic staffed by anesthesia nurses who are specialists in applying PVCs.
* Everyone will three times be asked to answer some questions in the DROP-IN, have their grip strength measured in both hands, and have the course of the veins in their arms clarified.
* The training group must do arm training exercises daily for at least eight weeks (training equipment is provided)
* Ten participants will at the end of the project period be invited to participate in a telephone interview about experiences of vein status during a cancer treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Planned neoadjuvant or adjuvant chemotherapy via intravenous peripheral venous cannula placed under ultrasound guidance
* PVC insertion is performed in the DROP-IN outpatient clinic, Department of Anesthesiology, Vejle Hospital, at least four times
* The patient has provided written and orally informed consent
* The patient must be cognitively well preserved and able to understand information

Exclusion Criteria:

* Patients who cannot read and understand Danish
* Patients <18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Level of pain as measure by the Numeric Rating Scale (score 1-10 where a low value defines low level of pain) | Measured at baseline
  Pain level after insertion of periphral venous catheter and at general activity measured with Numeric Rating Scale
Level of pain as measure by the Numeric Rating Scale (score 1-10 where a low value defines low level of pain) | Measured after five weeks of training/control
  Pain level after insertion of periphral venous catheter and at general activity measured with Numeric Rating Scale
Level of pain as measure by the Numeric Rating Scale (score 1-10 where a low value defines low level of pain) | Measured after eight weeks of training/control
  Pain level after insertion of periphral venous catheter and at general activity measured with Numeric Rating Scale

SECONDARY OUTCOMES:
Vein status | Measured at baseline
  Number of useable veins (assessed via ultrasound)
Vein status | Measured after five weeks of training/controll
  Number of useable veins (assessed via ultrasound)
Vein status | Measured after eight weeks of training/control
  Number of useable veins (assessed via ultrasound)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne I Jensen, PhD, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Southern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No